CLINICAL TRIAL: NCT01214343
Title: Randomized Controlled Trial Comparing Efficacy of Sorafenib Versus Sorafenib In Combination With Low Dose Cisplatin /Fluorouracil Hepatic Arterial InfUSion Chemotherapy in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Comparing Efficacy of Sorafenib Versus Sorafenib in Combination With Low-dose FP in Patients With Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Kinki University Faculty of Medicine, Department of Gastroenterology and Hepatology, Kinki University Faculty of Medicine, Department of Gastroenterology and Hepatology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SILIUS Phase III trial
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-10

CONDITIONS: Advanced Hepatocellular Carcinoma; Carcinoma; Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms
Keywords: sorafenib; Hepatic intraarterial infusion chemotherapy; HAIC; Low dose FP; cisplatin; fluorouracil
MeSH Terms: conditions — Carcinoma; Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib with Low-dose FP (Experimental)
  Interventions: Drug: Sorafenib with Low-dose FP
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib with Low-dose FP — Sorafenib will be administered orally at a dose of 400 mg bid for 28 days in a cycle. Cisplatin at the dose of 20 mg/m2 will be administered at day 1 and day8, and fluorouracil at the dose of 330 mg/m2 will be administered continuously at day 1-day 5, and day8-day12 via the implanted catheter system. A cycle is defined as 28 days.
  Other Names: Nexavar; Low-dose FP
  Arms: Sorafenib with Low-dose FP
Drug: Sorafenib — Sorafenib will be administered orally at a dose of 400 mg bid for 28 days in each cycle.A cycle is defined as 28 days.
  Other Names: Nexavar
  Arms: Sorafenib

SUMMARY:
The purpose of this study is to evaluate the efficacy of sorafenib in combination with low dose cisplatin /fluorouracil hepatic arterial infusion chemotherapy in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Sorafenib with Low-dose FP Group

Sorafenib will be administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid) for 28 days. Cisplatin at the dose of 20mg/m2 will be administered at day 1 and day8, and fluorouracil at the dose of 330mg/m2 will be administered continuously at day1-day5, and day8-day12 via the implanted catheter system.

Sorafenib Group

Sorafenib will be administered orally at a dose of 400 mg (2 x 200 mg tablets) twice daily (bid) for 28 days.

The treatment regimen will be continued until radiographic or symptomatic progression, the development of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. 20 Years and older.
2. Life expectancy of at least 12 weeks at the pre-treatment evaluation.
3. Advanced hepatocellular carcinoma with histological evidence on a biopsy specimen, or typical findings by dynamic CT or CT during hepatic arteriography/arterioportography.
4. Not suitable for resection or local ablation therapy or transcatheter arterial chemoembolization.
5. ECOG Performance status of 0 or 1.
6. Cirrhotic status of Child-Pugh score ≤ 7.
7. Adequate bone marrow, liver and renal function, as assessed by the following laboratory requirements:

   * Hemoglobin ≥8.5 g/dl
   * Granulocytes≥1500/μL
   * Platelet count ≥50,000 /μL
   * PT-INR ≤ 2.3
   * Total serum bilirubin ≤ 2 mg/dl
   * AST(SGOT) and ALT(SGPT) ≤ 6 × upper limit of normal
   * Serum creatinine ≤ 1.5 × upper limit of normal
   * Amylase ≤ 2 × upper limit of normal
8. Written Informed Consent must be obtained.

Exclusion Criteria:

1. Previous malignancy (except for cervical carcinoma in situ, adequate treated basal cell carcinoma, or superficial bladder tumors [Ta, Tis and T1], early gastric cancer, or other malignancies curatively treated > 3 years prior to entry
2. Renal failure
3. Any heart disease as follows

   * Congestive heart failure defined as NYHA class III or IV
   * Active coronary artery disease or ischemic heart disease such as cardiac infarction within 6 months prior to screening
   * Serious cardiac arrhythmia
   * Serious hypertension
4. Active clinically serious infections except for HBV and HCV
5. Active chicken pox.
6. Auditory disorder.
7. Known history of HIV infection.
8. Known metastatic or meningeal tumors.
9. Extrahepatic tumor spread which affects patient's prognosis
10. History of seizure disorder.
11. Clinically significant gastrointestinal bleeding within 4 weeks prior to study entry.
12. Embolization or infarction such as transient ischemic disease, deep vein thrombosis, pulmonary embolization.
13. Any history of treatment as follows:

    * Treatment with the agent which induces CYP3A4
    * Surgical procedure within 4 weeks prior to start of study drug
    * History of organ allograft
14. Patients unable to swallow oral medications.
15. Gastrointestinal disease that may affect to the absorption of drug or pharmacokinetics.
16. Medication that may affect to the absorption of drug or pharmacokinetics.
17. Any disease or disorder that may affect the evaluation of study drug.
18. Entry to the other clinical trial within 4 weeks prior to entry to this study.
19. Pregnant or breast-feeding patients.
20. Known allergy to the investigational agent or any agent given in association with this trial.
21. Substance abuse, medical, psychological or social conditions that, in the judgment of the investigator, is likely to interfere with the patient's participation in the study or evaluation of the stuy results.
22. Any condition that is unstable or could jeopardize the safety of the patient and its compliance in the study, in the investigator's judgment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Overall survival is defined as the time from randomization to death due to any cause

SECONDARY OUTCOMES:
Time to progression | TTP is defined as the time from randomization to radiological progression.
Progression Free Survival | PFS is defined as the time from randomization to radiological progression or death due to any cause
Change of tumor marker | Every 4-6 weeks
Biomarker predicting the efficacy | Pre and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Masatoshi Kudo, Professor, Study Chair — Kinki University Faculty of Medicine, Department of Gastroenterology and Hepatology
Locations (30):
- Japan (30):
  - Chiba University Hospital, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kurume University Medical Center, Kurume, Fukuoka
  - Gifu Municipal Hospital, Gifu, Gifu
  - Ogaki Municipal Hospital, Ōgaki, Gifu
  - Hiroshima City Hospital, Hiroshima, Hiroshima
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo Medical University, Sapporo, Hokkaido
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Japanese Red Cross Takamatsu Hospital, Takamatsu, Kagawa-ken
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Center for Gastroenterological and Hepatological Diseases, Miyazaki, Miyazaki
  - National Hospital Organization Nagasaki Medical Center, Ohmura, Nagasaki
  - Saiseikai Niigata Dai-ni Hospital, Niigata, Niigata
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Kawasaki Medical School Hospital, Kurashiki, Okayama-ken
  - Okayama University Hospital, Okayama, Okayama-ken
  - Ikeda Municipal Hospital, Ikeda, Osaka
  - Osaka Red Cross Hospital, Osaka, Osaka
  - Kinki University Hospital, Ōsaka-sayama, Osaka
  - Osaka University Hospital, Suita, Osaka
  - The University of Tokushima Faculty of Medicine, Tokushima, Tokushima
  - Kyorin University Hospital, Mitaka, Tokyo
  - Musashino Red Cross Hospital, Musashino, Tokyo
  - Juntendo University Nerima Hospital, Nerima City, Tokyo
  - Kyoundo Hospital, Tokyo, Tokyo
  - National Cancer Center Hospital, Tokyo, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi

REFERENCES:
- [Derived] Kudo M, Ueshima K, Yokosuka O, Ogasawara S, Obi S, Izumi N, Aikata H, Nagano H, Hatano E, Sasaki Y, Hino K, Kumada T, Yamamoto K, Imai Y, Iwadou S, Ogawa C, Okusaka T, Kanai F, Akazawa K, Yoshimura KI, Johnson P, Arai Y; SILIUS study group. Sorafenib plus low-dose cisplatin and fluorouracil hepatic arterial infusion chemotherapy versus sorafenib alone in patients with advanced hepatocellular carcinoma (SILIUS): a randomised, open label, phase 3 trial. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):424-432. doi: 10.1016/S2468-1253(18)30078-5. Epub 2018 Apr 7. PMID 29631810
- [Derived] Ueshima K, Kudo M, Tanaka M, Kumada T, Chung H, Hagiwara S, Inoue T, Yada N, Kitai S. Phase I/II Study of Sorafenib in Combination with Hepatic Arterial Infusion Chemotherapy Using Low-Dose Cisplatin and 5-Fluorouracil. Liver Cancer. 2015 Dec;4(4):263-73. doi: 10.1159/000367751. Epub 2015 Oct 21. PMID 26734580